CLINICAL TRIAL: NCT01432002
Title: Application of 18F-[FDG] PET/CT to Simulation and Planning of Radiotherapy (RT) for Breast Cancer. Definition of Target Volume for 3-D RT and for Partial Breast Irradiation (PBI) by IMRT Technique
Brief Title: FDG-PET/CT for Simulation and Radiation Treatment Planning of Early Breast Cancer
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Vincent Vinh-Hung, Privat Docent, University of Geneva, Switzerland
Other Study IDs: HUG 07-153
Record Dates: First submitted 2011-09-02; First posted 2011-09-12 (Estimated); Last update posted 2022-12-21 (Actual); Status verified 2022-12

CONDITIONS: Breast Neoplasm
Keywords: breast carcinoma; FDG; PET/CT; PET/IRM
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of the study is:

* to assess the potential benefits of 18F-[FDG] PET/CT and PET/MRI for operable breast cancer in order to define the size and location of the primary tumor, as well as axillary, supraclavicular and internal mammary lymph nodes.
* to apply the imaging results to the simulation and the radiation treatment planning and partial breast for 3-D radiation treatment and partial breast irradiation with intensity modulated radiation treatment (IMRT).

DETAILED DESCRIPTION:
Pre-operative FDG PET/CT, and in option PET/IRM, are intended for women with histologically confirmed operable clinically node-negative breast cancer, in whom breast conserving and post-operative radiotherapy are planned.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed breast carcinoma
* Clinical stage T1-2 N0 M0
* Age > 18 years
* Signed informed consent

Exclusion Criteria:

* WHO performance index 3
* Premenopausal women without contraception
* Gestation
* Lactating
* Prior surgery or radiotherapy on the same breast
* Unable to understand study participation
* Bilateral breast cancer
* Prior CT thorax-abdomen and breast MRI within 4 months of interview
* Presence of electromechanical implant and/or body ferromagnetic material
* Previous history of renal insufficiency requiring dialysis and/or hospitalisation
* Ureum and/or creatinine within 2 weeks of interview above lab's reference limits
* History of contrast allergy
* Hyperthyroidy
* Claustrophobia.

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women with operable clinically node-negative breast cancer
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2007-11; Primary Completion 2013-05 (Actual); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Drawing of target volumes | Up to 12 weeks after surgery
  Compare the drawing of target volumes using the PET/CT, PET/IRM information, or without these imaging informations.

SECONDARY OUTCOMES:
Correlate the FDG PET/CT PET/IRM with surgical pathology findings | Up to 12 weeks after surgery
  Compare the pre-operative imaging information with histopathological description of the resected primary tumor, and with the extent of lymph node involvement.

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Vinh-Hung, MD, PhD, Principal Investigator — Radiation Oncology, Geneva University Hospitals
Locations (1):
- Radiation oncology, Geneva University Hospitals, Geneva, Switzerland

REFERENCES:
- [Background] Bral S, Vinh-Hung V, Everaert H, De Coninck P, Storme G. The use of molecular imaging to evaluate radiation fields in the adjuvant setting of breast cancer: a feasibility study. Strahlenther Onkol. 2008 Feb;184(2):100-4. doi: 10.1007/s00066-008-1769-7. PMID 18259702
- [Background] Vinh-Hung V, Everaert H, Lamote J, Voordeckers M, van Parijs H, Vanhoeij M, Verfaillie G, Fontaine C, Vees H, Ratib O, Vlastos G, De Ridder M. Diagnostic and prognostic correlates of preoperative FDG PET for breast cancer. Eur J Nucl Med Mol Imaging. 2012 Oct;39(10):1618-27. doi: 10.1007/s00259-012-2181-1. Epub 2012 Jul 10. PMID 22777335
- [Background] Tabouret-Viaud C, Botsikas D, Delattre BM, Mainta I, Amzalag G, Rager O, Vinh-Hung V, Miralbell R, Ratib O. PET/MR in Breast Cancer. Semin Nucl Med. 2015 Jul;45(4):304-21. doi: 10.1053/j.semnuclmed.2015.03.003. PMID 26050658
- [Background] Vinh-Hung V, Everaert H, Gorobets O, Van Parijs H, Verfaillie G, Vanhoeij M, Storme G, Fontaine C, Lamote J, Perrin J, Farid K, Nguyen NP, Verschraegen C, De Ridder M. Breast cancer preoperative 18FDG-PET, overall survival prognostic separation compared with the lymph node ratio. Breast Cancer. 2021 Jul;28(4):956-968. doi: 10.1007/s12282-021-01234-z. Epub 2021 Mar 10. PMID 33689151
- [Background] Perrin J, Farid K, Van Parijs H, Gorobets O, Vinh-Hung V, Nguyen NP, Djassemi N, De Ridder M, Everaert H. Is there utility for fluorine-18-fluorodeoxyglucose positron-emission tomography scan before surgery in breast cancer? A 15-year overall survival analysis. World J Clin Oncol. 2022 Apr 24;13(4):287-302. doi: 10.5306/wjco.v13.i4.287. PMID 35582655